CLINICAL TRIAL: NCT01002261
Title: Determination of Hepatic Metabolism of Galactose and the Galactose Analog FDGal in Patients With Liver Disease and Healthy Subjects
Brief Title: Hepatic Metabolism of Galactose and the Galactose Analog FDGal in Patients With Liver Disease and Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Susanne Keiding (PI), Aarhus University Hospital, 8000 Aarhus C, Denmark
Other Study IDs: gal-FDGal; R01DK074419 (NIH)
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2009-10

CONDITIONS: Liver Cirrhosis
Keywords: Galactose; PET/CT; Liver physiology; Liver pathophysiology
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Liver cirrhosis / healthy subjects: 10 patients with liver cirrhosis and 10 sex and age-matched healthy subjects
- Liver cirrhosis and healthy subjects: Patients with liver cirrhosis and healthy subjects

SUMMARY:
The elimination of the carbohydrate galactose is used in daily clinical work with liver patients as a quantitative measure of metabolic liver function, as the liver test "The Galactose Elimination Capacity", GEC. We are working to develop a PET/CT scanning procedure for providing 3D images of the hepatic galactose elimination and measurement of regional values. This may be used for example for planning resection or stereotactic radiotherapy of a patient with malignant tumor in the liver. Will the patient be able to tolerate removal of the necessary part of the liver? We will include 10 patients with liver cirrhosis and 6 healthy human subjects. Direct measurements of the hepatic galactose elimination (successive constant iv infusions of galactose in increasing doses with measurements of blood concentrations of galactose in blood from an artery and a liver vein, and measurements of liver blood flow by indocyanine green, Ficks principle) are compared with PET/CT measurements after iv injection of a 18F-labelled galactose analog, FDGal.

Based on previous studies in pigs, we perform detailed calculations of the hepatic galactose elimination kinetics by the two methods, including estimation of a factor ("lumped constant") for recalculating PET/CT data to data for natural galactose.

Besides possible practical clinical importance, the project elucidates basic problems concerning liver metabolism using PET.

ELIGIBILITY:
Inclusion Criteria:

* liver cirrhosis

Exclusion Criteria:

* hepatic encephalopathy
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are out-patients recruited from Department of Hepatology, Aarhus University Hospital Healthy subjects are recruited via add in a local newspaper
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2009-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Lumped constant for recalculation of PET/CT data for FDGalactose to data for natural galactose | May 2011

CONTACTS AND LOCATIONS:
Overall Officials: John Westensee, Mr, Study Director — Research Support Office, Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, PET Centre, Aarhus, Denmark

REFERENCES:
- [Background] Sorensen M, Munk OL, Mortensen FV, Olsen AK, Bender D, Bass L, Keiding S. Hepatic uptake and metabolism of galactose can be quantified in vivo by 2-[18F]fluoro-2-deoxygalactose positron emission tomography. Am J Physiol Gastrointest Liver Physiol. 2008 Jul;295(1):G27-G36. doi: 10.1152/ajpgi.00004.2008. Epub 2008 May 15. PMID 18483186